CLINICAL TRIAL: NCT02004938
Title: Characteristics of the Internal Jugular Vein by Ultrasonography During Respiration in Children
Brief Title: Internal Jugular Ultrasound Measures During Respiration in Children
Status: Completed | Type: Observational
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Michelle D. Stevenson, Professor, University of Louisville
Other Study IDs: IRB 13.0345
Record Dates: First submitted 2013-08-19; First posted 2013-12-09 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Ultrasound Measurements; Normative Values
Keywords: measurements; jugular; ultrasound; pediatric; respiratory; diameter

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- normal respiratory function: This will include the 40 subjects enrolled in the study
  Interventions: Device: Sonosite Titan Ultrasound Machine

INTERVENTIONS:
Device: Sonosite Titan Ultrasound Machine

SUMMARY:
Project Aims: The purpose of this study is to determine the size of the right internal jugular vein (RIJV) in children with normal respiratory physiology during the respiratory cycle and evaluate the reliability of those measurements.

Hypothesis: Ultrasound measurements of internal jugular vein collapse of children can be reliably measured in the respiratory cycle.

Intervention: We will ensure that the patient is not having any respiratory symptoms or signs of dehydration. A clinical asthma score will be assigned using the Modified Woods pulmonary index scoring system. The Gorelick Dehydration Scale with also be calculated.

Using bedside ultrasonography with the Sonosite Titan ultrasound machine, each measurement will be taken with the subject lying in bed with the head of the bed elevated at 45 degrees with the subject's head in the neutral position and then turned 45 degrees leftward. Measurements of the internal jugular vein at maximal inhalation and exhalation will be recorded. Reliability calculations will be assessed.

ELIGIBILITY:
Inclusion Criteria:

Subjects ages 6-17 years old presenting to the emergency department (ED) will be enrolled into the normal respiratory function group.

Exclusion Criteria:

Children will be excluded from participation if they have: a baseline chronic lung disorder (including asthma), current respiratory illness, fever, Emergency Services Index (ESI) triage category of less than or equal to 2 (emergent acuity), chronic cough, dyspnea with exercise, wheezing, or a history of smoking by self and/or parent report.

Subjects will be excluded if they had prior cardiac/pulmonary disease or surgeries (other than asthma for the acute exacerbation group), significant musculoskeletal abnormalities (such as scoliosis) that might compromise baseline pulmonary function testing, a history of smoking tobacco or marijuana, and prematurity (birth at less than 37 weeks gestation. In addition, those with an allergy to ultrasound gel will be excluded from participation.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: pediatric emergency department
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Measurement of diameter of right internal jugular vein during the respiratory cycle at max inhalation and exhalation | During ED stay at initiation of intervention

SECONDARY OUTCOMES:
Clinical Asthma Score | During ED stay at initiation of intervention
  Will be recorded using Modified Woods pulmonary index scoring system.
Measurement of level of dehydration | During ED stay
  Will measure using the Gorelick scale.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle D Stevenson, MD, MS, Principal Investigator — University of Louisville
Locations (1):
- Kosair Children's Hospital, Louisville, Kentucky, United States